CLINICAL TRIAL: NCT00080990
Title: An Open-Labeled, Non-Randomized Phase I Study of Alvocidib (Flavopiridol) Administered With Oxaliplatin and Fluorouracil/Leucovorin in Patients With Advanced Solid Tumors
Brief Title: Alvocidib, Oxaliplatin, Fluorouracil, and Leucovorin Calcium in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00055; NCI-2009-00055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-03146; CDR0000357606; NCI-6365; 03-146A (Other: Memorial Sloan-Kettering Cancer Center); 6365 (Other: CTEP); U01CA069856 (NIH); NCT01645501 (obsolete NCT alias); NCT01664299 (obsolete NCT alias)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alvocidib; Fluorouracil; Oxaliplatin; Leucovorin

ARMS (1):
- Treatment (alvocidib with oxaliplatin, 5-FU, leucovorin) (Experimental): Patients receive alvocidib IV over 1 hour, oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 48 hours on days 1, 15, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, the cohort is expanded and an additional 10 patients are treated at that dose.
  Interventions: Drug: alvocidib; Drug: fluorouracil; Drug: oxaliplatin; Drug: leucovorin calcium

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV

SUMMARY:
This phase I trial is studying the side effects and best dose of alvocidib when given together with oxaliplatin, fluorouracil, and leucovorin calcium in treating patients with advanced solid tumors. Drugs used in chemotherapy, such as alvocidib, oxaliplatin, fluorouracil, and leucovorin calcium, work in different ways to stop tumor cells from dividing so they stop growing or die. Alvocidib may also make tumor cells more sensitive to chemotherapy. Combining more than one chemotherapy drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of flavopiridol when given in combination with oxaliplatin, fluorouracil, and leucovorin calcium in patients with advanced solid tumors.

II. Determine the pharmacokinetics of this regimen in these patients. III. Determine, preliminarily, the therapeutic activity of this regimen in these patients.

IV. Determine the dose-limiting toxicity and the recommended phase II dose of flavopiridol when administered with this regimen in these patients.

V. Determine the safety and tolerability of this regimen in these patients. VI. Correlate p21, p53, and apoptotic markers with response in patients treated with this regimen.

OUTLINE: This is a non-randomized, open-label, dose-escalation study of flavopiridol.

Patients receive alvocidib intravenously (IV) over 1 hour, oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 48 hours on days 1, 15, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of alvocidib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, the cohort is expanded and an additional 10 patients are treated at that dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor

  * Refractory to standard therapy or no standard therapy exists
* Evaluable disease
* No known untreated CNS metastases

  * Patients who have undergone local treatment for brain metastases and whose brain metastases are stable by repeat imaging study performed ≤ 4 weeks after treatment are allowed
* No primary CNS tumors
* Performance status - Karnofsky 60-100%
* WBC ≥ 3,500/mm^3
* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN for liver metastases)
* Creatinine ≤ 1.5 mg/dL
* No cardiac arrhythmias within the past 6 months
* No congestive heart failure within the past 6 months
* No myocardial infarction within the past 6 months
* No arterial or venous thrombosis within the past year
* No peripheral neuropathy > grade 1
* No other medical condition that would preclude study participation
* No serious or uncontrolled infection
* HIV negative
* Not pregnant or nursing

  * No nursing during and for 2 months after study participation
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation
* At least 2 weeks since prior immunotherapy
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin)
* No prior flavopiridol
* At least 2 weeks since prior radiotherapy
* Recovered from all prior therapy
* No concurrent therapy for thrombosis

  * Prophylaxis for central lines or deep vein thrombosis allowed
* No other concurrent investigational medications
* No concurrent vitamins, antioxidants, or herbal preparations and supplements

  * Concurrent single-tablet multivitamin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-02; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of biweekly alvocidib when given in conjunction with oxaliplatin, 5-fluorouracil, and leucovorin calcium | 6 weeks
  Defined as the dose level immediately preceding the dose where 2 or more patients experienced dose-limiting toxicity.

SECONDARY OUTCOMES:
Dose-limiting toxicity as defined by the occurrence of Grade 4 hematologic toxicity, Grade 3 or 4 non-hematologic toxicity including diarrhea despite antidiarrheal prophylaxis, or any delay in treatment resulting in less than 3 treatments in 6 weeks | 6 weeks
Recommended phase II dose of alvocidib | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Schwartz, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States